CLINICAL TRIAL: NCT01571960
Title: A Phase 1 Placebo Controlled Clinical Trial to Evaluate the Safety and Immunogenicity of a Prime-Boost Vaccine Regimen of GEO-D03 DNA and MVA/HIV62B Vaccines in Healthy, HIV-1-Uninfected Vaccinia Naive Adult Participants
Brief Title: Evaluating the Safety and Immune Response of a Prime-Boost HIV Vaccine Regimen in Healthy, HIV-Uninfected, Vaccinia-Naive Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: GeoVax, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 094; 11827 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1: study vaccine (Experimental): Participants in this arm will receive a 0.3-mg dose injection of GEO-D03 DNA vaccine at Days 0 and 56, followed by injections of MVA62B vaccine at Days 112, 168, and 224.
  Interventions: Biological: GEO-D03 DNA vaccine; Biological: MVA/HIV62B (MVA62B) vaccine
- Group 1: placebo vaccine (Placebo Comparator): Participants in this arm will receive injections of placebo for GEO-D03 DNA vaccine at Days 0 and 56, followed by injections of placebo for MVA62B vaccine at Days 112, 168, and 224.
  Interventions: Biological: Placebo for GEO-D03 DNA; Biological: Placebo for MVA62B:
- Group 2: study vaccine (Experimental): Participants in this arm will receive a 3-mg dose injection of GEO-D03 DNA vaccine at Days 0 and 56, followed by injections of MVA62B vaccine at Days 112, 168, and 303.
  Interventions: Biological: GEO-D03 DNA vaccine; Biological: MVA/HIV62B (MVA62B) vaccine
- Group 2: placebo vaccine (Placebo Comparator): Participants in this arm will receive injections of placebo for GEO-D03 DNA vaccine at Days 0 and 56, followed by injections of placebo for MVA62B vaccine at Days 112, 168, and 303.
  Interventions: Biological: Placebo for GEO-D03 DNA; Biological: Placebo for MVA62B:
- Group 3: study vaccine (Experimental): Participants in this arm will receive a 3-mg dose injection of GEO-D03 DNA vaccine at Days 0 and 56, followed by injections of MVA62B vaccine at Days 112 and 224.
  Interventions: Biological: GEO-D03 DNA vaccine; Biological: MVA/HIV62B (MVA62B) vaccine
- Group 3: placebo vaccine (Placebo Comparator): Participants in this arm will receive injections of placebo for GEO-D03 DNA vaccine at Days 0 and 56, followed by injections of placebo for MVA62B vaccine at Days 112 and 224.
  Interventions: Biological: Placebo for GEO-D03 DNA; Biological: Placebo for MVA62B:

INTERVENTIONS:
Biological: GEO-D03 DNA vaccine — Either a 0.3-mg (Group 1: study vaccine) or 3-mg dose (Groups 2 and 3: study vaccine) administered as a 1-mL IM injection into the deltoid
  Arms: Group 1: study vaccine; Group 2: study vaccine; Group 3: study vaccine
Biological: MVA/HIV62B (MVA62B) vaccine — 1 x 10^8-TCID50 dose of MVA62B vaccine, administered as a 1-mL IM injection into the deltoid
  Arms: Group 1: study vaccine; Group 2: study vaccine; Group 3: study vaccine
Biological: Placebo for GEO-D03 DNA — Administered as a 1-mL IM injection into the deltoid
  Arms: Group 1: placebo vaccine; Group 2: placebo vaccine; Group 3: placebo vaccine
Biological: Placebo for MVA62B: — Administered as a 1-mL IM injection into the deltoid
  Arms: Group 1: placebo vaccine; Group 2: placebo vaccine; Group 3: placebo vaccine

SUMMARY:
This study will test the safety and immune responses of a prime-boost regimen of two HIV vaccines- a DNA vaccine followed by a modified vaccinia Ankara (MVA) vaccine- in healthy, HIV-uninfected, vaccinia-naive adults.

DETAILED DESCRIPTION:
Although multiple candidate HIV vaccines are being studied, there is not yet an effective preventive HIV vaccine. This study will test the safety and immune responses of prime-boost regimens of two HIV vaccines: two injections of GEO-D03 DNA priming vaccine followed by either two or three boosting injections of MVA/HIV62B (MVA62B) vaccine.

This study will enroll 48 healthy, HIV-1-uninfected, vaccinia-naive adults into 1 of 3 groups. Participants within each group will be randomly assigned to receive either the study vaccine regimen (40 total participants) or placebo vaccine regimen (8 total participants).

The total study duration will be approximately 45 months. Participants in Group 1 will attend clinic visits for 14 months followed by annual health contacts, for a total of 3 years after initial study injection. Participants in Group 2 will attend clinic visits for 22 months followed by annual health contacts, for a total of 3 years after initial study injection. Participants in Group 3 will attend clinic visits for 20 months followed by annual health contacts, for a total of 3 years after initial study injection. Participants in Group 1 will have 17 study visits, participants in Group 2 will have 23 visits, and participants in Group 3 will have 21 visits.

At the screening visit, participants will give a medical history and undergo a complete physical exam, electrocardiogram (ECG), urine collection, blood collection, interview, HIV test, and pregnancy test (for participants who were born female). Participants will receive an intramuscular (IM) vaccination (study vaccine or placebo) into the deltoid on the schedule assigned to their group. The vaccination schedule is as follows: Group 1 participants will receive an injection on Days 0, 56, 112, 168, and 224; Group 2 participants will receive an injection on Days 0, 56, 112, 168, and 303; Group 3 participants will receive an injection on Days 0, 56, 112, and 224. On vaccination visits, participants will also undergo an abbreviated physical exam, a pregnancy test (for participants who were born female), risk-reduction counseling, and blood collection. Immediately following vaccination, participants will remain in the clinic for observation for 30 minutes; participants will be given a post-vaccination symptom log and instructed on how to complete it. Follow-up visits will consist of a brief physical exam, blood collection, and interview; some follow-up visits may also consist of a urine collection, HIV test, or ECG.

The last clinic visit will be at Day 425 for participants in Group 1, Day 667 for participants in Group 2, and Day 607 for participants in Group 3; after this visit, participants will be contacted for annual health follow-up consisting of confirming vital status, collecting safety information, and reporting a new HIV diagnosis or a pregnancy. A clinic visit will only be required if HIV confirmatory testing is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: participant demonstrates understanding of this study and completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks, amenable to HIV risk-reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years following initial study injection
* Agrees not to enroll in another study of an investigational research agent prior to completion of last required protocol clinic visit (excludes annual contacts for safety surveillance)
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Assessed by the clinic staff as being at low risk of HIV infection
* Hemoglobin greater than or equal to 11.0 g/dL for participants who were born female, or greater than or equal to 13.0 g/dL for participants who were born male
* White blood cell (WBC) count of 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelet level of 125,000 to 550,000/mm^3
* Chemistry panel: ALT, AST, alkaline phosphatase, and creatinine values less than or equal to institutional upper limits of normal
* Negative HIV-1 and HIV-2 blood test: U.S. participants must have a negative Food and Drug Administration (FDA)-approved immunoassay
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus (HCV) antibodies or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine: negative urine glucose, negative or trace urine protein, and negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis for red blood cells [RBCs] within institutional normal range)
* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
* Reproductive status: A participant who was born female must either: (1) Agree to consistently use effective contraception for sexual activity that could lead to pregnancy, from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using any of the following methods: condoms (male or female) with or without a spermicide, diaphragm or cervical cap with spermicide, intrauterine device (IUD), hormonal contraception, or successful vasectomy in the male partner (considered successful if a participant reports that a male partner has either documentation of azoospermia by microscopy or a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy); or (2) Not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation; or (3) Be sexually abstinent.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

* Vaccinia (smallpox) vaccine determined by (1) clinical evidence of vaccinia scarification; (2) self-reported history of vaccinia vaccination; (3) date of birth; or (4) U.S. military service prior to 1989 or after December 2002 (not excluded: a participant born before 1975, or with past U.S. military service, who self-reports he/she did not receive vaccinia vaccine and has no evidence of scarification)
* Untreated or incompletely treated syphilis infection
* HIV vaccine(s) received in a prior HIV vaccine trial. For potential participants who have received control/placebo in an HIV vaccine trial, the HVTN 094 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For potential participants who have received control/placebo in an experimental vaccine trial, the HVTN 094 PSRT will determine eligibility on a case-by-case basis. For potential participants who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 094 PSRT on a case-by-case basis.
* Immunosuppressive medications received within 168 days before first vaccination. Not excluded: (1) corticosteroid nasal spray for allergic rhinitis; (2) topical corticosteroids for mild, uncomplicated dermatitis; or (3) oral/parenteral corticosteroids given for non-chronic conditions not expected to recur (length of therapy 10 days or less with completion at least 30 days prior to enrollment)
* Blood products received within 120 days before first vaccination
* Immunoglobulin received within 60 days before first vaccination
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Investigational research agents received within 30 days before first vaccination
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 094 study
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response
  * A process that would require medication that affects the immune response
  * Any contraindication to repeated injections or blood draws
  * A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being during the study period
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine; or
  * Any condition specifically listed among the exclusion criteria below
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain (not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child)
* Hypersensitivity to eggs or egg products
* History of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up)
* ECG with clinically significant findings or features that would interfere with the assessment of myocarditis/pericarditis as determined by a contract ECG lab or cardiologist, including any of the following:

  * Conduction disturbance (complete left or complete right bundle branch block or nonspecific intraventricular conduction disturbance with QRS greater than or equal to 120 ms, PR interval greater than or equal to 220 ms, any second or third degree atrioventricular (AV) block, or QTc prolongation greater than 450 ms)
  * Repolarization (ST segment or T wave) abnormality that will interfere with the assessment of myocarditis/pericarditis
  * Significant atrial or ventricular arrhythmia
  * Frequent atrial or ventricular ectopy (e.g., frequent premature atrial contractions or two premature ventricular contractions in a row)
  * ST elevation consistent with ischemia; or
  * Evidence of past or evolving myocardial infarction
* Autoimmune disease
* Immunodeficiency
* Asthma other than mild, well-controlled asthma. Exclude a participant who:

  * Generally uses a bronchodilator (beta2 agonist) daily
  * In the past year, has any of the following:

    * More than one exacerbation of symptoms treated with oral steroids (note: oral/parenteral steroid use for asthma is exclusionary within 168 days before first vaccination)
    * Routinely used moderate to high dose inhaled corticosteroids (e.g., more than the equivalent of 250 mcg fluticasone, 400 mcg budesonide, 500 mcg beclomethasone, or 1,000 mcg triamcinolone/flunisolide, as a daily dose) or theophylline for asthma; or
    * Needed emergency care, urgent care, hospitalization, or intubation for asthma
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (not excluded: history of isolated gestational diabetes)
* Thyroidectomy or thyroid disease requiring medication during the last 12 months
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm mercury (Hg) systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings that must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these participants, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment
* Body mass index (BMI) greater than or equal to 40 or BMI greater than or equal to 35 with two or more of the following: age greater than 45, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, or known hyperlipidemia
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (not excluded: a participant with a surgical excision and subsequent observation period that in the investigator's estimation has a reasonable assurance of sustained cure or is unlikely to recur during the period of the study)
* Seizure disorder (not excluded: a participant with a history of seizures who has not required medications or had a seizure within the past 3 years)
* Asplenia: any condition resulting in the absence of a functional spleen
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are participants with psychoses within the past 3 years, ongoing risk of suicide, or history of suicide attempt or gesture within the past 3 years.
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04; Primary Completion 2014-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of local injection site reactogenicity signs and symptoms | Measured within the initial 72-hour period following each vaccination visit (Days 0, 56, 112, 168, 224, and 303)
  Signs and symptoms include pain, tenderness, erythema, induration, and maximum severity of pain and/or tenderness.
Frequency and severity of systemic reactogenicity signs and symptoms and maximum severity of systemic symptoms | Measured within the initial 72-hour period following each vaccination visit (Days 0, 56, 112, 168, 224, and 303)
  Systemic reactogenicity signs and symptoms include fever, malaise/fatigue, myalgia, headache, nausea, vomiting, chills, and arthralgia.
Distribution of values of safety laboratory measures: complete blood count (CBC), alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, and creatinine | Group 1: Measured through Day 334; Group 2: Measured through Day 394; Group 3: Measured through Day 334
Frequency of adverse events (AEs) categorized by MedDRA System Organ Class and MedDRA Preferred Term; severity and assessed relationship to study products; detailed description of all AEs meeting DAIDS criteria for expedited reporting | Group 1: Measured through Day 425; Group 2: Measured through Day 667; Group 3: Measured through Day 607
Report of the number of participants with early discontinuation of vaccinations, by treatment group and reason for discontinuation | Group 1: Measured through Day 425; Group 2: Measured through Day 667; Group 3: Measured through Day 607

SECONDARY OUTCOMES:
Frequency and magnitude of HIV-1 envelope (env)-specific binding antibody and isotypes | Group 2: Measured at Day 317; Group 3: Measured at Day 238
Frequency of neutralizing antibody responses to HIV-1 | Group 2: Measured at Day 317; Group 3: Measured at Day 238
In individuals with neutralizing antibodies to HIV-1, neutralizing antibody titers (magnitude) and breadth of neutralizing activity | Group 2: Measured at Day 317; Group 3: Measured at Day 238
Frequency and magnitude of HIV-1 specific CD4+ and CD8+ T cell responses as measured by intracellular cytokine staining (ICS) at 2 weeks after the second vaccination for Groups 2 and 3 | Measured at Day 70
Frequency and magnitude of HIV-1 specific CD4+ and CD8+ T cell responses as measured by ICS at 2 weeks after the last vaccination for Groups 2 and 3 | Group 2: Measured at Day 317; Group 3: Measured at Day 238
Avidity indices for env-specific binding antibody | Group 2: Measured at Day 317; Group 3: Measured at Day 238
Concentrations of secreted cytokines and chemokines by multiplex analysis of stimulated cell supernatants following peptide stimulation of PBMC 2 weeks after the last vaccination for Groups 2 and 3 | Group 2: Measured at Day 317; Group 3: Measured at Day 238
Blood concentrations of lymphocyte populations (T, B, and NK cells), dendritic cells, monocytes, and granulocytes | Measured through Day 126 (in Groups 2 and 3)
Concentrations of cytokines and chemokines in serum and/or plasma samples | Measured through Day 126 (in Groups 2 and 3)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Buchbinder, Study Chair — San Francisco Department of Public Health; Christine (Mhorag) Hay, Study Chair — University of Rochester
Locations (4):
- United States (4):
  - Alabama CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York

REFERENCES:
- [Background] Goepfert PA, Elizaga ML, Sato A, Qin L, Cardinali M, Hay CM, Hural J, DeRosa SC, DeFawe OD, Tomaras GD, Montefiori DC, Xu Y, Lai L, Kalams SA, Baden LR, Frey SE, Blattner WA, Wyatt LS, Moss B, Robinson HL; National Institute of Allergy and Infectious Diseases HIV Vaccine Trials Network. Phase 1 safety and immunogenicity testing of DNA and recombinant modified vaccinia Ankara vaccines expressing HIV-1 virus-like particles. J Infect Dis. 2011 Mar 1;203(5):610-9. doi: 10.1093/infdis/jiq105. Epub 2011 Jan 31. PMID 21282192
- [Background] Pantaleo G, Esteban M, Jacobs B, Tartaglia J. Poxvirus vector-based HIV vaccines. Curr Opin HIV AIDS. 2010 Sep;5(5):391-6. doi: 10.1097/COH.0b013e32833d1e87. PMID 20978379
- [Derived] Buchbinder SP, Grunenberg NA, Sanchez BJ, Seaton KE, Ferrari G, Moody MA, Frahm N, Montefiori DC, Hay CM, Goepfert PA, Baden LR, Robinson HL, Yu X, Gilbert PB, McElrath MJ, Huang Y, Tomaras GD; HIV Vaccine Trials Network (HVTN) 094 Study Group. Immunogenicity of a novel Clade B HIV-1 vaccine combination: Results of phase 1 randomized placebo controlled trial of an HIV-1 GM-CSF-expressing DNA prime with a modified vaccinia Ankara vaccine boost in healthy HIV-1 uninfected adults. PLoS One. 2017 Jul 20;12(7):e0179597. doi: 10.1371/journal.pone.0179597. eCollection 2017. PMID 28727817